CLINICAL TRIAL: NCT03381092
Title: Sentinel Lymph Node Biopsy in Clinically Node-negative Early Breast Cancer Patients After Neoadjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Director of Breast Center of Peking University Cancer Hospital, Peking University
Other Study IDs: BCP21
Record Dates: First submitted 2017-12-04; First posted 2017-12-21 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Invasive Breast Cancer
Keywords: neoadjuvant chemotherapy; sentinel lymph node biopsy; axillary lymph node dissection; Predictive model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Axillary lymph node status are determined in SLNB(sentinel lymph node biopsy) and surgical specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- invasive breast cancer: Patients with invasive breast cancer who have clinically negative axilla and receive neoadjuvant treatment followed by sentinel lymph node biopsy are eligible for this study.

SUMMARY:
This is a prospective, single-center, non-randomized, non-controlled observational study.

DETAILED DESCRIPTION:
The panel of the St. Gallen International Expert Consensus Conference on the Primary Therapy of Early Breast Cancer 2017 strongly believed that sentinel lymph node biopsy to be appropriate and favored the biopsy be carried out after neoadjuvant treatment in patients who presented with a clinically negative axilla and who received neoadjuvant treatment.

Patients with clinically node-negative early breast cancer treated in Breast Cancer Prevention and Treatment Center Peking University Cancer Hospital from February 2013 to August 2017 were retrospectively analyzed to investigate whether sentinel lymph node (SLN) biopsy after neoadjuvant chemotherapy can reduce the positive rate of SLN and the rate of axillary lymph node dissection (ALND). The study group underwent SLN biopsy after neoadjuvant chemotherapy, and the control group underwent SLN biopsy before chemotherapy. A total of 395 patients were eligible, including 85 in the study group and 310 in the control group. The detection rate of SLNs was 95.3% vs 98.7%（χ2 = 3.922，P = 0.069） in the study group compared with the control group, the positive rate of SLNs was 1.2% vs 18.6%（χ2 = 15.207，P = 0.000）, and the rate of ALND was 5.9% vs 15.2%（χ2 = 5.024，P = 0.025） in univariate analysis. Multivariate analysis showed that the study group had lower SLN positive rate (OR = 0.052, 95% CI: 0.0070 to 0.38, P = 0.004) and ALND rate (OR = 0.310, 95% CI: 0.118 to 0.812, P = 0.017). There was no statistically significant difference in detection rate of SLNs （OR = 0.244, 95% CI: 0.058 to 1.021, P = 0.053）between the two groups.

The aim of this study is to explore the detection rate and positive rate of sentinel lymph nodes, the rate of axillary lymph node dissection, and the proportion of patients with axillary lymph node metastases after neoadjuvant chemotherapy in patients with clinically node-negative early breast cancer. A mathematical model of axillary lymph node status will be established to predict axillary lymph node metastases.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer diagnosed with core needle needle biopsy;
* Staging cT1b-2N0M0;
* ER/PR positive cells ratio <10%, or HER2 positive (according to ASCO-CAP guidelines),and with chemotherapy indications;
* Without chemotherapy contraindications, and planned or has started neoadjuvant chemotherapy (HER2 positive breast cancer neoadjuvant anti-HER2 treatment, or have adjuvant anti-HER2 treatment plan);
* With axillary sentinel lymph node biopsy indications confirmed prior to neoadjuvant therapy;
* Voluntarily join the study and sign an informed consent form.

Exclusion Criteria:

* History of malignant tumors.
* With chemotherapy contraindications.
* Recieved any form of surgery of primary tumor or axillary lymph nodes.
* Refuse neoadjuvant chemotherapy.
* Refuse assessment examinations.
* Refuse to join the study.

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Invasive breast cancer patients with clinically negtive axilla.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Positive Rate of Axillary Sentinel Lymph Nodes. | Within 6 weeks after obtaining the post-surgery pathological results.
  Positive rate of axillary sentinel lymph nodes in patients with clinically node-negative early breast cancer after neoadjuvant chemotherapy will be assessed.

SECONDARY OUTCOMES:
Detection Rate of Axillary Sentinel Lymph Nodes. | Within 6 weeks after obtaining the post-surgery pathological results.
  Detection rate of axillary sentinel lymph nodes in patients with clinically node-negative early breast cancer after neoadjuvant chemotherapy will be assessed.
Rate of Axillary Lymph Node Dissection. | Within 6 weeks after obtaining the post-surgery pathological results.
  Rate of axillary lymph node dissection in patients with clinically node-negative early breast cancer after neoadjuvant chemotherapy will be assessed.
Proportion of Patients with Axillary Lymph Node Metastases. | Within 6 weeks after obtaining the post-surgery pathological results.
  Proportion of patients with axillary lymph node metastases in patients with clinically node-negative early breast cancer after neoadjuvant chemotherapy will be assessed.
Axillary Lymph Nodes Status Prediction Model. | Within 6 weeks after obtaining the post-surgery pathological results.
  A mathematical model of axillary lymph node status will be established to predict axillary lymph node metastases in patients with early stage axillary cancer after neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Qi-jun Zheng, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China